CLINICAL TRIAL: NCT07335042
Title: Development of an Interpretable Prediction Model for Myocardial Injury After Noncardiac Surgery in Patients Undergoing Major Hepatobiliary Surgery
Brief Title: Prediction Model for MINS After Major Hepatobiliary Surgery
Status: Recruiting | Type: Observational
Sponsor: Beijing Tsinghua Chang Gung Hospital (Other)
Responsible Party: Principal Investigator, Zhifeng Gao, Associate Professor, Beijing Tsinghua Chang Gung Hospital
Other Study IDs: 25454-4-01-01
Record Dates: First submitted 2026-01-04; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Myocardial Injury After Noncardiac Surgery (MINS); Postoperative Complications; Liver Neoplasm; Hepatobiliary Diseases
Keywords: MINS; Major Hepatobiliary Surgery; Hepatectomy; Hepatic Inflow Occlusion; Pringle Maneuver; Prediction Model; High-sensitivity Cardiac Troponin
MeSH Terms: conditions — Postoperative Complications; Liver Neoplasms; Digestive System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Cohort: Adult patients scheduled for major hepatobiliary surgery at Beijing Tsinghua Chang Gung Hospital and other participating centers.
  Interventions: Procedure: Major Hepatobiliary Surgery

INTERVENTIONS:
Procedure: Major Hepatobiliary Surgery — Patients undergo standard major hepatobiliary surgery (e.g., hepatectomy). The specific surgical strategy, including the method of hepatic inflow occlusion (e.g., Pringle maneuver or SPVO), is determined by the attending surgeon based on routine clinical practice and patient condition, not by the study protocol.

SUMMARY:
This multi-center, prospective observational study aims to develop and validate an interpretable prediction model for Myocardial Injury After Noncardiac Surgery (MINS) in patients undergoing major hepatobiliary surgery. The study adopts a nested modeling strategy, starting with baseline risk factors (e.g., RCRI) and stepwise incorporating hepatic inflow occlusion strategies (specifically comparing SPVO vs. Pringle maneuver) and routine intraoperative biomarkers. The model's performance will be evaluated using AUC, Net Reclassification Improvement (NRI), and Decision Curve Analysis (DCA), followed by interpretability analysis using SHAP values and external validation in an independent cohort.

DETAILED DESCRIPTION:
Study Design and Methodology: The study consists of four consecutive phases aimed at constructing a robust and interpretable prediction model for MINS.

1. Multi-center Cohort Standardization: Based on clinical data from multiple participating centers, the investigators will establish a standardized structural dataset. Strict inclusion and exclusion criteria will be applied. The process involves rigorous data cleaning and normalization to harmonize demographics, surgical operation details, and perioperative hemodynamic parameters across different centers, laying the foundation for model construction.
2. Nested Modeling and Performance Evaluation: A nested modeling strategy will be employed to assess the incremental predictive value of specific surgical and biological variables:

   Model A (Baseline): Constructed using standard baseline variables such as the Revised Cardiac Risk Index (RCRI).

   Model B (+Surgical Technique): Incorporates hepatic inflow occlusion strategies, specifically comparing SPVO (Selective Pringle Vascular Occlusion) vs. Pringle maneuver, along with occlusion duration and frequency.

   Model C (Full Model): Further incorporates MINS-related biomarkers.

   Model performance will be comprehensively evaluated using:

   Discrimination: Area Under the Receiver Operating Characteristic Curve (AUC).

   Calibration: Calibration plots.

   Clinical Utility: Net Reclassification Improvement (NRI) and Decision Curve Analysis (DCA) to assess the improvement in risk stratification and clinical net benefit after adding new variables.
3. Model Interpretability Analysis: To enhance the transparency of the model ("White-box" approach), SHAP (SHapley Additive exPlanations) values or similar methods will be utilized. This will quantify and visualize the specific contribution (weight) of key variables, such as SPVO usage, to the individual risk prediction, aligning the statistical results with clinical medical reasoning.
4. External Validation: The final model will undergo validation using an independent external clinical cohort. This step aims to test the stability and generalizability of the model across different center data, defining its applicable scope in real-world clinical scenarios.

ELIGIBILITY:
Inclusion Criteria:

Adults (18-85 yr, ASA physical status II-III) undergoing major hepatobiliary surgery were enrolled. Major surgery was defined as duration ≥ 3 h involving hepatectomy (≥ 3 segments) or biliary reconstruction necessitating ICU admission. Eligibility required paired perioperative high-sensitivity cardiac troponin T (hs-cTnT) data and comprehensive documentation of surgical covariates, including surgical approach (laparoscopic vs. open), resection nature (anatomic vs. non-anatomic), number of resected segments, tumor characteristics (size and location), and presence of cirrhosis.

Exclusion Criteria:

(1) preoperative acute myocardial infarction, unstable angina, heart failure, or chronic kidney disease (estimated glomerular filtration rate < 60 ml/ (min · 1.73 m2); (2) undocumented inflow occlusion strategy; or (3) non-imputable missing covariates.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1800
Sampling Method: Non-Probability Sample
Enrollment: 1800 (Estimated)
Dates: Start 2025-06-11 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Myocardial Injury After Noncardiac Surgery | Within 30 days after surgery
  MINS is defined as myocardial injury resulting from myocardial ischemia (that may or may not result in necrosis) occurring within 30 days after surgery.
  The diagnosis is based on a peak high-sensitivity cardiac troponin (hs-cTn) level exceeding the 99th percentile upper reference limit (URL) due to presumed ischemic etiology, irrespective of the presence of ischemic symptoms or electrocardiographic (ECG) changes.
  Routine hs-cTn screening will be performed on postoperative days 1, 2, and 3. Additional measurements will be taken if clinical signs of ischemia occur anytime within the 30-day follow-up period.

SECONDARY OUTCOMES:
30-day All-cause Mortality | Within 30 days after surgery
  Death from any cause postoperatively.
Postoperative Length of Hospital Stay | Up to 90 days
  Duration from surgery to hospital discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Zhifeng Gao, MD, Principal Investigator — Beijing Tsinghua Changgeng Hospital
Locations (6):
- China (6):
  - Beijing Tsinghua Changgung Hospital, School of Clinical Medicine, Tsinghua Medicine，Tsinghua University, Beijing
  - Peking University International Hospital, Beijing
  - The First Affiliated Hospital of Army Medical University, Chongqing
  - Qingdao West Coast New Area People's Hospital, Qingdao
  - The First Affiliated Hospital of Shandong First Medical University, Shandong
  - Zhuhai People's Hospital, Zhuhai

IPD SHARING:
Plan to Share IPD: Undecided